CLINICAL TRIAL: NCT06924489
Title: Effect of 3-Dimensional Imaging Device on Advanced Adenoma Detection During Colonoscopy: A Multi-center Randomized Controlled Trial
Brief Title: Advanced Adenoma Detection With 3D Imaging Device During Colonoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Beijing Friendship Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KY20242132-F-1
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Adenoma; Colorectal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2D imaging arm (Active Comparator): participants will undergo colonoscopy examination using 2D imaging colonoscope
  Interventions: Procedure: Colonoscopy after bowel cleansing with 2D imaging device
- 3D imaging arm (Experimental): participants will undergo colonoscopy examination using 3D imaging colonoscope
  Interventions: Procedure: Colonoscopy after bowel cleansing with 3D imaging device

INTERVENTIONS:
Procedure: Colonoscopy after bowel cleansing with 2D imaging device — participants will undergo colonoscopy examination using 2D imaging colonoscope to detect potential adenomas or polyps. The classification of the detected lession will be determined by the edoscopic diagnosis based on the JNET classification system or by the pathological diagnosis with tissues from biopsy or polypectomy.
  Arms: 2D imaging arm
Procedure: Colonoscopy after bowel cleansing with 3D imaging device — participants will undergo colonoscopy examination using 3D imaging colonoscope to detect potential adenomas or polyps. The classification of the detected lession will be determined by the edoscopic diagnosis based on the JNET classification system or by the pathological diagnosis with tissues from biopsy or polypectomy.
  Arms: 3D imaging arm

SUMMARY:
The goal of this clinical trial is to learn if 3-dimensional (3D) imaging device works to identify patients with high risk adenomas during colonoscopy to guide proper follow-up strategy. It will also learn about the safety of 3-dimensional (3D) imaging device. The main questions it aims to answer are:

Does 3-dimensional (3D) imaging device improve the identification of patients with high risk adenomas? What adverse events do participants experience during colonoscopy? Researchers will compare 3-dimensional (3D) imaging device to traditional 2-dimensional (2D) imaging device to see if 3-dimensional (3D) imaging device works to improve high risk adenoma identification.

Participants will:

Undertake colonoscopy examination using 3-dimensional (3D) imaging device or 2-dimensional (2D) imaging device. Be followed-up to 30 days to record potential colonoscopy-relevant adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* Patients with indications for colonoscopy and receiving diagnostic colonoscopy, without history of inflammatory bowel disease, colorectal cancer, polypectomy or polyposis syndromes;
* Signing the written informed consent;

Exclusion Criteria:

* Patients with polyposis syndromes (e.g., Peutz-Jeghers syndrome, Cronkhite-Canada syndrome, familial adenomatous polyposis [FAP], Lynch syndrome, etc.);
* Patients with a history of colorectal polypectomy and pathological diagnosed as adenoma;
* Patients with a history of colorectal adenocarcinoma or alarming symptoms;
* Patients with a history of inflammatory bowel disease;
* Patients with mental illness or severe functional disorder who cannot cooperate with colonoscopy;
* Patients with severe cardiopulmonary insufficiency;
* Patients with severe coagulation disorders or high bleeding risk (platelets <50×10⁹/L, INR >1.5; discontinuation of antithrombotic drugs should follow the 2012 Japanese Guidelines for Gastroenterological Endoscopy in Patients Undergoing Antithrombotic Treatment and the2017 Appendix on Anticoagulants Including Direct Oral Anticoagulants;
* Patients with severe electrolyte imbalances;
* Patients with acute peritonitis or suspected intestinal perforation;
* Patients with toxic megacolon;
* Patients with stage 3 or higher hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg);
* Patients with untreated severe abdominal hernia, intestinal obstruction;
* Patients with intestinal strictures of any cause;
* Pregnancy and lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1566 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
High-risk adenoma (HRA) detection rate | 1-7 days after polypectomy
  HRA were defined with one of the following features:1. diameter ≥10 mm or 2. (tubulo)villous adenomas or 3. with high-grade dysplasia or 4. sessile serrated lesions (SSLs) or 5. ≥ 3 adenomas. SSLs were defined as lesions with at least one crypt showing a characteristic sessile serrated lesion-type appearance.
  HRA detection rate is defined as the number of participants diagnosed with HRA divided by the total number of participants

SECONDARY OUTCOMES:
Adenoma detection rate (ADR) | 1-7 days after polypectomy
  The number of participants with at least 1 adenoma divided by the total number of participants
Polyp detection rate (PDR) | 1-7 days after polypectomy
  The number of participants with at least 1 polyp divided by the total number of participants
Clinically relevant serrated polyp detection rate | 1-7 days after polypectomy
  Clinically relevant serrated polyps are defined as ≥10 mm serrated polyps (SPs, including hyperplastic polyps, SSLs, and traditional serrated adenomas) and >5 mm SPs in the proximal colon.
  Clinically relevant serrated polyp detection rate is defined as the number of participants with at least 1 clinically relevant serrated polyp divided by the total number of participants.
Modified advanced adenoma detection rate | 1-7 days after polypectomy
  Modified advanced adenoma are defined with one of the following features:1. diameter ≥10 mm or 2. (tubulo)villous adenomas or 3. with high-grade dysplasia or 4. sessile serrated lesions (SSLs). SSLs were defined as lesions with at least one crypt showing a characteristic sessile serrated lesion-type appearance.
  Modified advanced adenoma detection rate is defined as the number of participants diagnosed with modified advanced adenoma divided by the total number of participants
Advanced adenocarcinoma detection rate | 1-7 days after polypectomy
  Advanced adenocarcinoma is defined as adenocarcinoma with submucosal invasion more than 1000μm (SM2). Advanced adenocarcinoma detection rate is defined as the number of participants diagnosed with advanced adenocarcinoma divided by the total number of participants
The number of lesions per colonoscopy | 1-7 days after polypectomy
  The number of lesions per colonoscopy was defined as the number of corresponding lesions (adenoma, polyp, clinically relevant serrated polyps, et al)divided by the total number of colonoscopies or participants
Lesion detection rate in different location | 1-7 days after polypectomy
  Lesion (adenoma, polyp, clinically relevant serrated polyps) detection rate in different location of colon and rectum
Lesion detection rate in different size | 1-7 days after polypectomy
  Lesion (adenoma, polyp, clinically relevant serrated polyps) detection rate in different size (≤3mm, 3-10mm, >10mm)
Lesion detection rate in different type | 1-7 days after polypectomy
  Lesion (adenoma, polyp, clinically relevant serrated polyps) detection rate in different type (Paris classification)
Lesion detection rate by endoscopists of different experience | 1-7 days after polypectomy
  Lesion (adenoma, polyp, clinically relevant serrated polyps) detection rate by endoscopists of different experience (senior or junior)
Cecal intubation time | immediately during the colonoscopy examination procedure
  Cecal intubation time (CIT) is defined as the time from the insertion of the colonoscope tip into the anal verge until reaching the cecal base or cecal end
Withdrawal time | immediately during the colonoscopy examination procedure
  Withdrawal time is defined as the time from reaching the cecal base or cecal end to the endoscope withdrawal to the anal verge, excluding the time of polypectomy
The colonoscopy-relevant adverse events | 1-30 days after polypectomy
  Aspiration pneumonia, perforation, bleeding, splenic injury/rupture, death, or others requiring hospitalization within 30 days after the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, M.D, Principal Investigator — Xijing Hospital of Digestive Disease

IPD SHARING:
Plan to Share IPD: No